CLINICAL TRIAL: NCT06006546
Title: 426c.Mod.Core-C4b Adjuvanted With 3M-052-AF + Alum Immunization in Combination With an Antiretroviral Analytical Treatment Interruption (ATI) in People Living With HIV for Elicitation of VRC01-lineage Antibodies
Brief Title: The Study of Immunization in People Living With HIV Undergoing an ATI for Elicitation of VRC01-lineage Antibodies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 807
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Chronic HIV Infection
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (ATI) (Experimental): Group 1 will receive 2 doses of the vaccine at Week 0 and 12. Group 1 will transition to Schedule 2 at the Week 14 visit. The Schedule 2 "ATI with Monitoring" phase can last for 24 weeks OR until any antiretroviral therapy (ART) re-initiation criteria are met, OR the ATI can continue longer with the approval of the Protocol Safety Review Team (PSRT) and the participant's primary HIV healthcare provider. Group 1 will transition to Schedule 3, the "Follow-up on ART restart" phase that lasts until study week 64, regardless of the point where it begins.
  Interventions: Biological: 426c.Mod.Core-C4b; Other: Adjuvant 3M-052-AF+Alum
- Group 2 (No ATI) Control (Experimental): Group 2 transitions from Schedule 1 into Schedule 4, "Follow-up on ART," at the Week 14 visit, and remains on Schedule 4 through study week 64.
  Interventions: Biological: 426c.Mod.Core-C4b; Other: Adjuvant 3M-052-AF+Alum

INTERVENTIONS:
Biological: 426c.Mod.Core-C4b — 100 mcg and 300 mcg
Other: Adjuvant 3M-052-AF+Alum — 5 mcg

SUMMARY:
This is a multicenter controlled interventional trial. This phase 1 trial is the first study to assess 426c.Mod.Core-C4b adjuvanted with 3M-052-AF + aluminum hydroxide suspension (Alum) in people living with HIV (PLWH).

DETAILED DESCRIPTION:
The aim of this study is to combine the ability of germline (GL)-targeting HIV-1 Envelope protein (Env)-derived immunogens to activate naïve B cells that express the unmutated GL forms of VRC01-class broadly neutralizing antibodies (bnAbs) with the booster capabilities of viral Envs that are expected to circulate in persons living with chronic HIV. The goals are: 1) to elicit VRC01-class GL and intermediate stage antibody responses in PLWH; 2) to identify the viral Envs that guided the maturation of the GL-VRC01 responses elicited by the GL-targeting Env immunogen; 3) during the time when viremia is detectable, the investigator will assess the stage of maturation of these VRC01 antibodies and if they affect viral replication; and 4) investigate how the virus may evolve to escape the activity of these antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to complete the informed consent process, including an Assessment of Understanding (AoU): Volunteer demonstrates an understanding of this study and completes a questionnaire prior to first vaccination with verbal demonstration of understanding of questionnaire items that were answered incorrectly.
2. 18 to 55 years old, inclusive, on day of enrollment.
3. Confirmed HIV infection as documented by medical records or confirmatory HIV testing at screening.
4. On suppressive ART for at least 48 weeks prior to screening. ART is defined as a combination therapy regimen including at least 1 integrase inhibitor and 1 nucleoside reverse transcriptase inhibitor (such as Dovato™) or 2 nucleoside reverse transcriptase inhibitors plus integrase inhibitors. Changes in ARVs for reasons other than virologic failure (eg, tolerability, simplification, different formulation, drug-drug interaction profile) are allowed within 48 weeks prior to screening and up until 6 weeks prior to screening. A fully active alternative ARV regimen is available, in the opinion of the Investigator, in the event of discontinuation of the current ARV regimen with development of resistance.
5. Plasma HIV RNA < 50 copies/mL (or lower limit of quantitation [LLOQ]) for at least 48 weeks prior to enrollment. NOTE: At least one viral load measurement within 48 weeks prior to the screening visit and another viral load from the screening prior to enrollment visit must be available for review. Two "blips" (ie, plasma HIV-1 RNA > LLOQ and < 400 copies/mL) are allowed if each blip is preceded and followed by values < LLOQ and if the blip(s) occur(s) more than 24 weeks prior to enrollment.
6. CD4+ cell count > 450 cells/mm3 and CD4+ cell % ≥ 15% obtained within 40 days prior to enrollment.
7. Available for clinic follow-up through the last clinic visit, willing to undergo leukapheresis, and willing to be contacted 12 months after the last study-product administration.
8. Agrees not to enroll in another study of an investigational agent during participation in the trial. If a potential participant is already enrolled in another clinical trial, approvals from the other trial sponsor and the HVTN 807 PSRT are required prior to enrollment into HVTN 807.
9. In good general health according to the clinical judgment of the site investigator.
10. Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator.
11. Total serum calcium of ≥ 8.5 mg/dL.
12. Hemoglobin (Hgb):

    * ≥ 10.0 g/dL for volunteers who were assigned female sex at birth (AFAB)
    * ≥ 11.0 g/dL for cisgender volunteers who were assigned male sex at birth (AMAB) and for transgender men who have been on hormone therapy for more than 6 consecutive months
    * ≥ 11.0 g/dL for transgender women who have been on hormone therapy for more than 6 consecutive months
    * For transgender volunteers who have been on hormone therapy for less than 6 consecutive months, determine Hgb eligibility based on their sex assigned at birth.
13. Absolute neutrophil count (ANC) ≥ 750/mm3

    .
14. Platelets ≥ 100,000/mm3

    .
15. Alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) based on the institutional normal range and direct bilirubin within the institutional range of normal.
16. Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73m2 as calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation.
17. For Group 1 volunteers: must agree to consistently use condoms from study week 14 through until viral load post-ATI is undetectable (at a minimum 20 weeks on study, at a maximum 64 weeks on study).
18. For Group 1 volunteers

    * Persons of pregnancy potential

      * Must have a negative beta human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on day of enrollment.
      * Must agree to use effective means of contraception from at least 21 days prior to enrollment until at least 8 weeks post last vaccination and viral load post-ATI is undetectable (at a minimum 20 weeks on study, at a maximum 64 weeks on study).
    * Volunteers who are AFAB or intersex at birth must agree to not seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization from at least 21 days prior to enrollment through until viral load post-ATI is undetectable (at a minimum 20 weeks on study, at a maximum 64 weeks on study).
19. For Group 2 volunteers

    * Persons of pregnancy potential:

      * Must have a negative β-HCG pregnancy test (urine or serum) on day of enrollment.
      * Must agree to use effective means of contraception from at least 21 days prior to enrollment until 8 weeks after their last scheduled vaccination (study week 20).
    * Volunteers who are AFAB or intersex at birth must agree to not seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.

Exclusion Criteria:

1. Current receipt of ART other than nucleoside reverse transcriptase inhibitor and integrase inhibitor.
2. Receipt of long-acting ART within 3 months of enrollment.
3. Documented history of resistance to any components of the current ARV regimen.
4. Known resistance to 1 or more drugs in 2 or more ARV drug classes. NOTE: M184V/I is an exception and should not be considered when assessing this criterion. Prior HIV resistance testing is not required.
5. ART initiation during acute HIV-1 infection (defined as within 1 year of HIV-1 acquisition, if known).
6. History of an HIV-associated malignancy (including Kaposi's sarcoma), and any type of lymphoma or virus-associated cancers.
7. History of HIV-associated neurocognitive disease or progressive multifocal leukoencephalopathy.
8. History of HIV-related illness under US Centers for Disease Control (CDC) Category C (except for recurrent pneumonia) within 10 years prior to screening, based on available medical history and assessed by the Investigator for clinical relevance. Anyone with a history of CD4 < 200 cells/mm3 on one or more occasions, based on available medical history and assessed by the Investigator for clinical relevance. Documentation of every case with history of CD4 < 200 cells/mm3 must be provided to the Sponsor and PSRT, who will determine eligibility on a case-by-case basis. NOTE: History of treated and resolved pulmonary tuberculosis (TB) will not be exclusionary.
9. Active or recent non-HIV-associated malignancy requiring systemic chemotherapy or surgery within 36 months prior to enrollment or for whom such therapies are expected in the subsequent 12 months. NOTE: Minor surgical removal of localized skin cancers (squamous cell carcinoma, basal cell carcinoma) is not exclusionary.
10. Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg), hepatitis C antibody without documented history of prior treatment and clearance, or hepatitis C virus RNA (HCV-RNA) in blood.
11. Diagnosis of cirrhosis.
12. Current untreated or incompletely treated active TB disease or untreated latent TB infection. NOTE: Individuals who are on treatment for latent TB with at least 4 weeks of treatment completed are not excluded.
13. Volunteer who is breastfeeding or pregnant.
14. Body mass index (BMI) ≥ 40. Enrollment of individuals with BMI ≥ 40, whom the site investigator assesses are in good health, may be considered by PSRT approval.
15. Diabetes mellitus (DM). Type 2 DM controlled with diet alone (and confirmed by HgbA1c ≤ 8% within the last 6 months) or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with Type 2 DM that is well controlled on hypoglycemic agent(s) may be considered by the PSRT on a case-by-case basis
16. History of or current clinical atherosclerotic cardiovascular disease (ASCVD), as defined by 2013 American College of Cardiology/American Heart Association (ACC/AHA) guidelines, including a previous diagnosis of any of the following:

    * Acute myocardial infarction
    * Acute coronary syndromes
    * Stable or unstable angina
    * Coronary or other arterial revascularization
    * Stroke
    * Transient ischemic attack
    * Peripheral arterial disease presumed to be of atherosclerotic origin
17. Previous or current recipient of an investigational HIV vaccine (previous placebo/control recipients are not excluded).
18. Receipt of non-HIV experimental vaccine(s) received within the last 1 year. Exceptions include vaccines that have subsequently undergone licensure or Emergency Use Authorization (EUA) by the FDA or World Health Organization (WHO) emergency use listing (EUL), or if outside the US, by the national Regulatory Authority (RA) authorizing this clinical trial.
19. Congenital or acquired immunodeficiency, including systemic medication use likely to impair immune response to vaccine in the opinion of the site investigator, such as history of systemic corticosteroids (long-term use), immunosuppressive anti-cancer or other immunosuppressive agents, interleukins, systemic interferons, systemic chemotherapy, or other medications considered significant by the investigator within the 24 weeks prior. Note: HIV is not exclusionary.
20. Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
21. Previous receipt of any anti-HIV monoclonal antibody.
22. Receipt of any of the following vaccines within 4 weeks prior to enrollment:

    * Live replicating vaccines
    * Any mRNA-based vaccine with FDA licensure, FDA EUA, or WHO EUL
    * ACAM2000 vaccine > 30 days prior with a vaccination scab still present.
23. Receipt of any vaccines that are not covered in #22 above within 14 days prior to enrollment. Please note this includes replication incompetent vaccines such as the Jynneos vaccine for the prevention of mpox (formerly known as monkeypox) disease.
24. Initiation of antigen-based immunotherapy (AIT) for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval. Note: Any AIT should be scheduled at least 14 days prior to enrollment.
25. Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life of greater than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
26. History of serious reaction (eg, hypersensitivity, anaphylaxis) to any vaccine or component of the study vaccine, including imidazoquinolone (eg, imiquimod).
27. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
28. Idiopathic urticaria within the past year.
29. Bleeding disorder diagnosed by a clinician which would make study procedures a contraindication (eg, factor deficiency, coagulopathy, platelet disorder requiring special precautions).
30. Seizure disorder; febrile seizures as a child or seizures secondary to alcohol withdrawal more than 5 years ago are not exclusionary.
31. Asplenia or functional asplenia.
32. Active duty and reserve US military personnel.
33. Any other chronic or clinically significant condition that, in the clinical judgment of the investigator, would jeopardize the safety or rights of the study participant, including but not limited to: clinically significant forms of substance use or alcohol use disorder(s), serious psychiatric disorders, persons with any suicide attempt within the past 1 year (if between 1 and 2 years, consult PSRT for approval), or cancer that, in the clinical judgement of the site investigator, has potential for recurrence (excluding basal cell carcinoma).
34. A participant with a history of a potential immune-mediated medical condition (PIMMC), either active or remote. Specific examples are listed in Appendix I (AESI Index). Not exclusionary: 1) Remote history of Bell's palsy (> 2 years ago) not associated with other neurologic symptoms and 2) mild psoriasis that does not require ongoing systemic treatment.
35. Investigator concern for difficulty with venous access based on clinical history and physical examination. For example, persons with a history of intravenous drug use or substantial difficulty with previous blood draws.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-10-27 (Estimated); Study Completion 2026-10-27 (Estimated)

PRIMARY OUTCOMES:
The number of participants local reactogenicity signs and symptoms | 14 days following each vaccination
The number of participants systemic reactogenicity signs and symptoms | 14 days following each vaccination
Number and description of serious adverse events (SAEs) | 12 months following any receipt of study product
  adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult AEs
Number and description of medically attended adverse events (MAAEs) | 12 months following any receipt of study product
  adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult AEs
Number and description of adverse events of special interest (AESIs) | 12 months following any receipt of study product
  adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult AEs
Number and description of AEs leading to early participant withdrawal or permanent discontinuation and reason for withdrawal/discontinuation | 12 months following any receipt of study product
  adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult AEs
Frequency of total Env-specific and CD4-bs-specific B cells, prior to ATI | At baseline (week 0) and after each vaccination
  as assessed by flow cytometry at baseline and after each vaccination
Frequency of VRC01-class BCR sequences of isolated CD4-bs B cells, prior to ATI | At baseline (week 0) and after each vaccination
  , as assessed by B-cell sorting and BCR sequencing
Frequency of Env-specific and CD4-bs-specific B cells | After week 16
  as assessed by flow cytometry
Frequency of VRC01-class BCR sequences of isolated CD4-bs B cells | After week 16
  as assessed by B-cell sorting and BCR sequencing

SECONDARY OUTCOMES:
Compare Env sequences during ATI in Group 1 participants that initiated the development of VRC01 antibodies and those that did not | Study duration or 12 months following any receipt of study product
Magnitude of Binding of selected recEnvs from Group 1 participants that initiated the development of VRC01-class antibodies to VRC01-class precursor and intermediate antibodies | Study duration or 12 months following any receipt of study product
Magnitude of Binding of selected recEnvs from Group 1 participants that initiated the development of VRC01-class antibodies to B cells expressing VRC01-class BCRs. | Study duration or 12 months following any receipt of study product

OTHER OUTCOMES:
Magntidue of binding and neutralizing activity of any VRC01-class antibodies isolated during the study | Study duration or 12 months following any receipt of study product
Frequency of occurrence of similarities s in viral sequences of Group 2 participants (if any viruses emerge on study) with Group 1 participants | Study duration or 12 months following any receipt of study product
Magnitude of participant and potential participant motivations, perceptions and tolerance for ATIs, for prolonged viremia, and for trial requirements (eg, ART switches, barrier protection for all sexual activity) | Study duration or 12 months following any receipt of study product
Magnitude of social benefits (eg, altruism) and negative social impacts, including but not limited to anxiety regarding being off ART and becoming viremic again and fear of inadvertent HIV transmission to partners | Study duration or 12 months following any receipt of study product
Magnitude of participant and potential participant decision-making quality, including perception of being informed, clarity and support in decision making, and satisfaction with their choice regarding participation. | Study duration or 12 months following any receipt of study product
Response rate of immunogenicity of each vaccine regimen, additional virologic and immunogenicity assays may be performed in a subset of participants, including on samples from other timepoints | Study duration or 12 months following any receipt of study product
Conduct analysis related to furthering the understanding of HIV, immunology, vaccines, and clinical trial conduct | Study duration or 12 months following any receipt of study product

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Birmingham, Birmingham, Alabama
  - Atlanta- Ponce, Atlanta, Georgia
  - The Hope Clinic of the Emory Vaccine Center CRS (Site #31440), Decatur, Georgia
  - BIDMC, Boston, Massachusetts
  - Columbia P&S CRS Site#30329, New York, New York
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - Seattle Vaccine and Prevention CRS (Site # 30331), Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No